CLINICAL TRIAL: NCT06966115
Title: Optimising Access to Vocational Rehabilitation Through Multiple Sclerosis Charities: A Feasibility Randomised Controlled Trial
Brief Title: Optimising Access to Vocational Rehabilitation for People With Multiple Sclerosis
Acronym: MS_Work_Hub
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Blanca de Dios Perez, Principal Investigator, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMHS 102-0325; 184 (Other Grant/Funding Number: UK MS Society)
Record Dates: First submitted 2025-04-24; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: Vocational Rehabilitation; multiple sclerosis; job retention
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSVR (Experimental): Participants in the MSVR group will be asked to complete a questionnaire booklet to explore variables of interest.
  Participants will then be invited to an optional semi-structured, feedback interview to provide qualitative information on their experience of the intervention.
  Interventions: Behavioral: Multiple Sclerosis Vocational Rehabilitation (MSVR)
- Control Group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Multiple Sclerosis Vocational Rehabilitation (MSVR) — MSVR involves an initial assessment (including vocational goal setting), followed by up to 10 hours of individually tailored support over six months according to need. The support will focus on supporting the person with MS to remain at work by addressing topics such as:
  * Understanding MS
  * Advice on reasonable adjustments
  * Support requesting reasonable adjustments
  * Fatigue management
  * Managing cognition at work
  * Information about legal rights
  * Disclosure
  * Long-term career planning
  * Managing mood difficulties
  * Signposting to local and national resources. MSVR addresses the individual needs of the person with MS and offers advice remotely (e.g., via telephone, videoconference, or email). The sessions will be arranged at a time convenient for the person, and the support needed will vary according to the complexity of their workplace difficulties.
  Arms: MSVR

SUMMARY:
People with multiple sclerosis (MS) often leave the workforce prematurely due to MS symptoms and difficulties managing workplace relationships and performance. Vocational rehabilitation (VR) can improve job retention outcomes for people with MS, but there is a lack of evidence on the effectiveness of these interventions.

A psychologist and occupational therapist-delivered VR intervention was previously developed to support people with MS to remain in paid employment. This programme was tested in a community setting and within the UK National Health Service (NHS). The preliminary findings demonstrate that the intervention is highly acceptable to people with MS and their employers and helped participants with MS to meet their vocational goals. However, the study also identified various barriers (e.g., lack of staff, service structure, etc.) to delivering this programme more widely within a healthcare setting.

Because of this, patient and public involvement (PPI) representatives suggested testing the VR intervention within the services provided by MS charities. This approach could be beneficial to reach people with MS who might be in the earlier stages of the illness and looking for information or who have not considered discussing "work" with their healthcare providers.

Therefore, the VR intervention MSVR ("multiple sclerosis vocational rehabilitation") was adapted to be delivered by non-specialists working for MS charities. Over recent years, the practice of training non-specialists to deliver evidence-based and complex interventions has increased to reach communities where there is a lack of resources or to help increase the reach of these interventions.

This study aims to:

1. Explore the feasibility and acceptability of providing employment support through MS charities.
2. Determine the parameters for a future large-scale randomised controlled trial.
3. Explore the experiences of those receiving and delivering the MSVR intervention.

Sixty people with MS in paid employment will be recruited to receive support with employment tailored to their needs over six months. Participants with MS will be asked to complete a booklet of questionnaires with variables known to affect employment status.

Approximately 20 participants will be asked to participate in a feedback interview at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18
2. Can give informed consent,
3. Can communicate in English,
4. Are in paid employment (including self-employed).

Exclusion Criteria:

1. Planning to retire within the next 12 months.
2. Currently receiving vocational rehabilitation support from the NHS or other employer services.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | At baseline, and -6, -9 and 12-months post-randomisation.
  The short form 36 health survey questionnaire measures eight health constructs relating to physical and mental health. The scale ranges from 0-100, with 100 representing highest level of health and functioning, and lower scores representing higher levels of disability. This measure has a high internal consistency (Cronbach's alpha >0.80) and good test-retest reliability (>0.70).
Work Productivity and Activity Impairment Questionnaire- Multiple Sclerosis | At baseline, and -6, -9 and 12-months post-randomisation.
  This questionnaire includes questions about the employment situation of the person with MS, hours missed at work due to MS, and two numerical scales measuring how MS impacts productivity at work and conducting everyday activities.
  The numeric scales range from 0 (no impact) to 10 (unable to perform an activity), where a higher score represents a larger impact of MS at work and conducting everyday life activities.
  The recall will be extended from seven days to four weeks.

SECONDARY OUTCOMES:
Goal Attaiment Scaling | At baseline, and -6, -9 and 12-months post-randomisation.
  The Goal Attainment Scale (GAS) (Turner-Stokes L., 2009) will be used to ascertain the intervention's impact on the vocational goals.
  Participants will be asked to evaluate whether or not they met the intervention goals using a 5-point scale from -2 (goal not met, much worse than expected) to +2 (goal met, much more than expected). A GAS T score will be calculated using the standardised formula for goal attainment. Goals are considered met if the GAS T score is >50.
Patient Health Questionnaire - 9 (PHQ-9) | At baseline, and -6, -9 and 12-months post-randomisation.
  Change in the level of depression symptoms. Higher scores indicate a worse outcome, total scores range from 0-27, scale values range from 0-3.
Generalised Anxiety Disorder - 7 (GAD-7) | At baseline, and -6, -9 and 12-months post-randomisation.
  Change in the level of anxiety symptoms. Higher scores indicate a worse outcome, total scores range from 0-21, scale values range from 0-3.
Perceived Difficulties Questionnaire | At baseline, and -6, -9 and 12-months post-randomisation.
  The Perceived Deficits Questionnaire (PDQ) (Sullivan et al. 1990) explores the perceived cognitive difficulties and measures four sub-scales within the questionnaire: attention/concentration, planning/organisation, retrospective memory and prospective memory.
  The PDQ is a 20-item scale scored with a 5-point Likert scale ranging from 0 (never) to 4 (almost always). The total score for the scale ranges between 0- 80 points, and the domain sub-scales range from 0-20; where a higher score represents a greater perceived cognitive deficits. There is no cut-off score for the sub-scales, but a score of ≥40 on the PDQ is considered as being in a "risk range".
Health-related quality of life | At baseline, and -6, -9 and 12-months post-randomisation.
  EQ-5D-5L - Five scaled questions assess five domains of quality of life (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each response corresponds to a 1-digit number. The total responses are combined into a 5-digit number to represent the health state; e.g., 11111 represents no problems in the health state. These are then converted to an index score; higher scores indicate greater health-related quality of life.
Fatigue levels | At baseline, and -6, -9 and 12-months post-randomisation.
  Modified Impact Fatigue Scale - 5 items (MFIS-5) (Fisk et al., 1994; Fischer et al., 1999). Total score ranges from 0-20; higher scores indicate greater impact of fatigue.
  Scale scores range from 0-4 with 5 scaled questions.
Self-efficacy | At baseline, and -6, -9 and 12-months post-randomisation.
  The Generalised Self-Efficacy Scale (GSE) assesses the participants' belief in their ability to complete tasks successfully. This scale has high internal consistency with alphas are between .76 and .90). The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Reasonable Adjustments | At baseline, and -6, -9 and 12-months post-randomisation.
  Questions regarding whether the employer has provided or not reasonable adjustments to the employee in the workplace.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Dios Perez B, Kendrick D, das Nair R, Evangelou N, Newsome I, Radford K. Optimising access to vocational rehabilitation through multiple sclerosis charities: Protocol for a feasibility randomised controlled trial. PLoS One. 2025 Jun 27;20(6):e0325570. doi: 10.1371/journal.pone.0325570. eCollection 2025. PMID 40577335